CLINICAL TRIAL: NCT03437577
Title: Comparison of the Cognitive and Motor Effects of Treatment Between an Immediate- and Extended-release Tacrolimus (Envarsus® XR) Based Immunosuppression Regimen in Kidney Transplant Recipients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PHARM-2017-25529
Record Dates: First submitted 2018-02-12; First posted 2018-02-19 (Actual); Results first posted 2021-04-15 (Actual); Last update posted 2021-04-15 (Actual); Status verified 2021-03

CONDITIONS: Kidney Transplant Failure and Rejection
Keywords: Kidney; Transplant
MeSH Terms: conditions — Rejection, Psychology | interventions — Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- immediate-release tacrolimus (Active Comparator): This is standard of care
  Interventions: Drug: immediate-release tacrolimus
- extended release tacrolimus (Experimental): replace standard of care
  Interventions: Drug: extended release tacrolimus

INTERVENTIONS:
Drug: immediate-release tacrolimus — Standard of care for transplant patients
  Other Names: Prograf
  Arms: immediate-release tacrolimus
Drug: extended release tacrolimus — Experimental care
  Other Names: Envarsus®XR.
  Arms: extended release tacrolimus

SUMMARY:
The primary objective is to compare the effect of treatment with an immediate-release tacrolimus to an extended-release tacrolimus (i.e., Envarsus® XR) immunosuppressive regimen on cognitive and motor function in kidney transplant recipients

DETAILED DESCRIPTION:
Between four (4) months and 14 months after receiving a kidney transplant and, per standard of care (SOC), having been placed on an immediate-release (IR) tacrolimus immunosuppressant regimen, participants in this study will undergo cognitive and motor function testing and have a blood sample collected (BASELINE). Half of the participants will then be randomly converted to extended-release (XR) tacrolimus (Envarsus® XR) while the other half will remain on IR tacrolimus for the duration of the study. Both the IR and XR groups will repeat the cognitive and motor function testing and have a blood sample collected at 6, 12, and 24 weeks Post-BASELINE. A practice version of the cognitive and motor function tests will be administered no more than 60 days prior to the baseline visit (Pre-BASELINE). Alternate versions of the cognitive and motor tests will be used at each Post-BASELINE testing session to control for possible practice effects.

The primary objective is to compare the effect of treatment with an immediate-release tacrolimus to an extended-release tacrolimus (i.e., Envarsus® XR) immunosuppressive regimen on cognitive and motor function in kidney transplant recipients.

The secondary objective is to determine the factors that explain inter-individual variability in cognitive response. Pharmacokinetic and demographic factors will be explored. Variability in cognitive response between individuals can be large. A population approach (nonlinear, mixed effects) will be used. Measurement of drug concentration will be the dependent variable.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female kidney transplant recipient;
2. 18-65 years of age;
3. receiving a kidney transplant from a living or deceased donor;
4. if female, premenopausal and heterosexually active, must be using two forms of highly effective birth control (at least one of which must be a barrier method) which includes consistent and correct usage of established oral contraception, established intrauterine device or intrauterine system, or barrier methods of contraception: condom or occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/suppository, starting at screening and throughout the study period and for 90 days after the final study drug administration;
5. written informed consent to participate in the study

Exclusion Criteria:

1. younger than 18 years of age;
2. older than 65 years of age;
3. Non-native level English speaker;
4. pregnant women
5. breastfeeding women

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2018-05-08 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan Marino, PhD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Extended-Release Tacrolimus: replace standard of care
  extended release tacrolimus: Experimental care
- Non-Randomized: Participants in this arm were not randomized to either arm. They ended study participation prior to randomization.
Period: Pre-Randomization
Arm/Group | Immediate-Release Tacrolimus | Extended-Release Tacrolimus | Non-Randomized
Started | 0 | 0 | 10
Completed | 0 | 0 | 0
Not Completed | 0 | 0 | 10
Not completed — Withdrawal by Subject | 0 | 0 | 10
Period: Post-Randomization
Arm/Group | Immediate-Release Tacrolimus | Extended-Release Tacrolimus | Non-Randomized
Started | 3 | 5 | 0
Completed | 3 | 3 | 0
Not Completed | 0 | 2 | 0
Not completed — Physician Decision | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Population: All participants are included at baseline, including those who withdrew participant prior to randomization
Groups:
- Total: Total of all reporting groups
Arm/Group | Immediate-Release Tacrolimus | Extended-Release Tacrolimus | Non-Randomized | Total
Number analyzed (Participants) | 3 | 5 | 10 | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 5 | 10 | 18
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.3 (9.5) | 60.4 (1.9) | 49.2 (10) | 52.8 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4 | 8
  Male | 1 | 3 | 6 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 1
  Asian | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 2 | 1 | 3
  White | 2 | 3 | 8 | 13
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 | 5 | 10 | 18

OUTCOME MEASURES:

1. Primary Outcome: Change in Controlled Oral Word Association Test (COWAT)
Description: During The Controlled Oral Word Association Test (COWAT), participants are asked to make verbal associations to different letters of the alphabet by saying all the words which they can think of beginning with a given letter. Three letters of progressively increasing associative difficulty are presented with 60 seconds allotted per letter for word retrieval. Scores are calculated as a sum of the total words produced across the 3 letter trials. The lowest possible score is zero, meaning no words could be produced. There is no limit to the higher end of the scale given that participants can produce as many words as possible for each of the three letters. Higher scores indicate greater word retrieval and better cognitive function. Outcome is reported as the change in COWAT between baseline and 6 weeks, baseline and 12 weeks, and baseline and 24 weeks.
Time Frame: Change from baseline at 6,12, 24 weeks
Population: All participants who were randomized and participated in outcome measure data collection are included.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Immediate-Release Tacrolimus | Extended-Release Tacrolimus
Number analyzed (Participants) | 3 | 5
score on a scale
  Baseline to 6 weeks | .44 (.51) | -2.11 (2.83)
  Baseline to 12 weeks | -0.88 (1.89) | -1.78 (2.01)
  Basline to 24 weeks | 0.78 (.84) | -0.44 (2.04)

ADVERSE EVENTS:
Time Frame: 24 weeks
Arm/Group | Immediate-Release Tacrolimus | Extended-Release Tacrolimus
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/5
Other Adverse Events (participants affected / at risk) | 0/3 | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-09-06): https://cdn.clinicaltrials.gov/large-docs/77/NCT03437577/Prot_SAP_000.pdf
  • Informed Consent Form (2018-04-26): https://cdn.clinicaltrials.gov/large-docs/77/NCT03437577/ICF_001.pdf